CLINICAL TRIAL: NCT03129932
Title: Effects Gluten on Body Composition, Energy Expenditure and Adipokine Profile in Non-celiac Women With Obesity
Brief Title: Effects Gluten Intake on Body Composition, Energy Expenditure and Adipokine Profile in Non-celiac Women With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacqueline Isaura Alvarez Leite (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor-Investigator, Jacqueline Isaura Alvarez Leite, MD.Ph.D; Full Professor, Federal University of Minas Gerais
Organization: Federal University of Minas Gerais (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 49480215.0.0000.5149
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Obesity
Keywords: gluten; adipokine; obesity; diet
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: double-masked, crossover, randomized, controlled study
Who Masked: Participant, Investigator
Masking Description: volunteers will receive placebo or gluten corn muffins that are similar in taste and appearance. Investigator does not know who is receiving placebo or gluten muffins. During analyses, each sample is coded to avoid volunteer or phase identification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gluten phase (Active Comparator): volunteers will receive 2 corn muffins containing12g of gluten/muffin to be consumed daily for 4 weeks
  Interventions: Dietary Supplement: gluten phase
- Placebo phase (Placebo Comparator): volunteers will receive 2 corn muffins without gluten/muffin to be consumed daily for 4 weeks
  Interventions: Dietary Supplement: placebo phase

INTERVENTIONS:
Dietary Supplement: gluten phase — 2 cakes containing 9g of vital gluten/each will be consume during the 4 weeks of intervention
  Arms: gluten phase
Dietary Supplement: placebo phase — 2 cakes without gluten will be consume during the 4 weeks of intervention
  Arms: Placebo phase

SUMMARY:
This is a double-masked, crossover, randomized, controlled study that aims to evaluate, in women with obesity, a possible influence of wheat gluten on food choices, body weight, resting metabolism and circulating inflammation markers and adipokines. The volunteers will be randomized into two groups, half of them will initiate the experiment by taking 2 placebo muffins daily for 4 weeks (Placebo phase) and the remnant volunteers will take 2 corn muffins containing 12g of gluten/each for 4 weeks (Gluten phase). At the 1st, 4th and 8th experimental weeks will be evaluated body weight, body composition, lipid profile, glucose, insulin, leptin, adiponectin, and inflammatory markers.

DETAILED DESCRIPTION:
It is a double-masked, crossover, randomized, controlled study. For this, volunteers will be kept on gluten-free diet for 8 weeks. At the first moment, a structured Food Frequency Questionnaire will be applied, as well as a 72-hour food register, to evaluate routine of food consumption and daily intake of gluten. The volunteers will be randomized into two groups, half of them will initiate the experiment by taking 2 placebo muffins daily for 4 weeks (Placebo phase) and the remnant volunteers will take 2 corn muffins containing 12g of gluten/each for 4 weeks (Gluten phase). After that, volunteers will be transferred for the other phase for 4 more weeks. During the 8 experimental weeks, all volunteers will be instructed to exclude any food containing gluten from their diet. At the 1st, 4th and 8th experimental weeks after 12 hours of fasting and 30 minutes of resting, volunteers will be submitted to indirect calorimetry, electrical bioimpedance, blood collection and anthropometry (weight and height). The volunteers will also respond a questionnaire about life habits, family history, previous history, physical activity and food frequency. Blood samples will be used to assess blood count, lipid profile, glucose, insulin, leptin, adiponectin, and inflammatory markers (soluble VCAM, C-reactive protein, fibrinogen). Four weeks after the end of the experiment, and return to the alimentary routine, body weight, blood sample, calorimetry and bioimpedance will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* Women between 20 and 50 years without diagnosis of celiac disease
* overweight and obese, respectively, BMI of 24.9- 34.9
* without menopause

Exclusion Criteria:

- Subjects with positive serology for celiac disease or allergy to wheat

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01-10 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in body Weight | 1st, 4th and 8th weeks
  measured in scale presented in kg

SECONDARY OUTCOMES:
Height | 1st week
  measured in meters
Changes in BMI | 1st, 4th and 8th weeks
  calculated by body weigh / square of height
Changes in resting metabolic rate | 1st, 4th and 8th weeks
  measured by indirect calorimetry in kcal/kg or kcal/day
Changes in macronutrient intake | 1st, 4th and 8th weeks
  calculation of food intake based on 24h diary - result in % kcal
waist circumference | 1st, 4th and 8th weeks
  measured in cm
Changes in IL-6 blood concentration | 1st, 4th and 8th weeks
  measure by ELISA in ug/mL
Changes in IL-10 | 1st, 4th and 8th weeks
  blood concentration measure by ELISA in ug/mL
Changes in IL-1beta | 1st, 4th and 8th weeks4th and 8th weeks
  blood concentration measure by ELISA in ug/mL
Changes in Adiponectin | 1st, 4th and 8th weeks
  blood concentration measure by ELISA in ug/mL
Changes in Leptin | 1st, 4th and 8th weeks
  blood concentration measure by ELISA in ug/mL
Changes in C reactive protein | 1st, 4th and 8th weeks
  blood concentration measure in mg/mL

CONTACTS AND LOCATIONS:
Overall Officials: JAQUELINE I ALVAREZ-LEITE, MD, PhD, Principal Investigator — Federal University of Minas Gerais

IPD SHARING:
Plan to Share IPD: No